CLINICAL TRIAL: NCT06379880
Title: Impact on Quality of Life and Health of the CONTINUUM+ CONNECT Remote Monitoring Solution: Prospective, Randomized, Multicenter Trial FEGALA
Brief Title: Impact on Quality of Life and Health of the CONTINUUM+ CONNECT Remote Monitoring Solution
Acronym: FEGALA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Paul Strauss (Other)
Collaborators: Continuum Plus Santé (Unknown); Plateforme nationale qualité de vie et cancer (Unknown); WeShare (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-031; 2024-A00120-47 (Other: ID-RCB Number)
Record Dates: First submitted 2024-04-11; First posted 2024-04-23 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Prostatic Neoplasms; Lung Neoplasms; Breast Neoplasms; Colorectal Neoplasms
Keywords: Remote patient monitoring; Metastatic cancer
MeSH Terms: conditions — Prostatic Neoplasms; Lung Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients using CONTINUUM+ CONNECT remote monitoring solution (Experimental)
  Interventions: Device: CONTINUUM+ CONNECT remote monitoring
- Patients with conventional follow-up without remote monitoring application. (No Intervention)

INTERVENTIONS:
Device: CONTINUUM+ CONNECT remote monitoring — CONTINUUM+ CONNECT is a web platform, accessible via the internet, which contains the digital medical device (DMN) Continuum+ alert module. This is a medical software intended for the interpretation of clinical constants, symptoms, adverse events and pain, generating alerts with a view to improving the monitoring of patients undergoing anticancer treatment. The "Continuum+ Alert Module" version 1.0.0 dated 30 April 2021 is CE-marked and will be used in accordance with the manufacturer's instructions for use by patients in the experimental group.
  Arms: Patients using CONTINUUM+ CONNECT remote monitoring solution

SUMMARY:
FEGALA is a comparative, multicenter, randomized, prospective, open-label study comparing the results observed at 3 months (± 15 days) on the EORTC QLQ-C30 scale in a group of patients with metastatic cancer followed on an outpatient basis and benefiting from the CONTINUUM+ CONNECT solution (with or without nursing support at home) versus comparable patients benefiting from conventional monitoring.

DETAILED DESCRIPTION:
CONTINUUM+ CONNECT is a platform, accessible from a computer, a smartphone or a tablet, allowing remote monitoring of cancer patients followed on an outpatient basis. The remotely monitored patient is invited to answer questionnaires (regarding adverse events, physiological constants and pain) at home. These questionnaires are either completed by the patient himself, if his condition allows it (self-assessment) or completed with the help of a professional on an outpatient basis (hetero-assessment). The data and alerts are transmitted in real time to the healthcare professionals in charge of the patient who analyze them and then determine the course of action to take.

In order to evaluate the impact of remote monitoring by CONTINUUM+ CONNECT on the quality of life and health of patients with metastatic cancer, the present prospective randomized multicenter study will be carried out.

Four main types of cancer will be studied: Breast, Lung, Colorectal and Prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged ≥ 18 years with a solid tumor (only breast, lung, colorectal, prostate cancer) at the metastatic stage followed on an outpatient basis;
2. Patients initiating oral and/or injectable anticancer treatment, whatever the line of treatment, administered on an outpatient basis including day hospitalization;
3. Patients who have given their written, free and informed consent;
4. Patients with life expectancy of more than 3 months;
5. Patients able to complete questionnaires according to the investigator's judgment, and to use the CONTINUUM+ CONNECT electronic application either alone or accompanied by a professional (home nurse);
6. Patients affiliated to a social security scheme or beneficiaries of such a scheme.

Exclusion Criteria:

1. Patients receiving home hospitalization care or being hospitalized at the time of treatment initiation;
2. Patients receiving concomitant radiotherapy;
3. Patients using another remote monitoring application;
4. Patients enrolled in another clinical trial;
5. Patients protected by law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2025-11-07 (Actual); Study Completion 2026-01-26 (Actual)

PRIMARY OUTCOMES:
Effect of the CONTINUUM+ CONNECT solution on the results in terms of physical health on the EORTC QLQ-C30 questionnaire in patients with metastatic cancer followed in outpatient settings who did not require assistance in self-assessment | At 3 months (± 15 days) post-inclusion
  Difference in physical health score from EORTC QLQ-C30 questionnaire at 3 months (± 15 days) in patients with metastatic cancer depending on intervention group

SECONDARY OUTCOMES:
Effect of CONTINUUM+ CONNECT solution on the results at 3 months (± 15 days) post-inclusion in terms of physical health on the EORTC QLQ-C30 questionnaire in patients with metastatic cancer followed in outpatient settings | At 3 months (± 15 days) post-inclusion
  Difference in physical health score from EORTC QLQ-C30 questionnaire at 3 months (± 15 days) in patients with metastatic cancer depending on intervention group (patients using CONTINUUM+ CONNECT solution (hetero- and self-assessment) or with conventional care)
Effect of CONTINUUM+ CONNECT solution on all dimensions of EORTC QLQ-C30 questionnaires (at 3 months) | At 3 months (± 15 days) post-inclusion
  Difference according to intervention group regarding all dimensions of EORTC QLQ-C30 questionnaires
Effect of CONTINUUM+ CONNECT solution on all dimensions of EORTC QLQ-C30 questionnaires (at 6 months) | At 6 months (± 15 days) post-inclusion
  Difference according to intervention group regarding all dimensions of EORTC QLQ-C30 questionnaires
Effect of the solution on specific symptom scales depending on the tumor localization (at 3 months) - breast cancer group | At 3 months (± 15 days) post-inclusion
  Difference on specific symptom scales QLQ-BR23
Effect of the solution on specific symptom scales depending on the tumor localization (at 3 months) - lung cancer group | At 3 months (± 15 days) post-inclusion
  Difference on specific symptom scales QLQ-LC13
Effect of the solution on specific symptom scales depending on the tumor localization (at 3 months) - prostate cancer group | At 3 months (± 15 days) post-inclusion
  Difference on specific symptom scales QLQ-PR25
Effect of the solution on specific symptom scales depending on the tumor localization (at 3 months) - colorectal cancer group | At 3 months (± 15 days) post-inclusion
  Difference on specific symptom scales QLQ-CR29
Effect of the solution on specific symptom scales depending on the tumor localization (at 6 months) - breast cancer group | At 6 months (± 15 days) post-inclusion
  Difference on specific symptom scales QLQ-BR23
Effect of the solution on specific symptom scales depending on the tumor localization (at 6 months) - lung cancer group | At 6 months (± 15 days) post-inclusion
  Difference on specific symptom scales QLQ-LC13
Effect of the solution on specific symptom scales depending on the tumor localization (at 6 months) - prostate cancer group | At 6 months (± 15 days) post-inclusion
  Difference on specific symptom scales QLQ-PR25
Effect of the solution on specific symptom scales depending on the tumor localization (at 6 months) - colorectal cancer group | At 6 months (± 15 days) post-inclusion
  Difference on specific symptom scales QLQ-CR29
Frequency of grade 3 - 4 adverse events present at 3 months post-inclusion | At 3 months (± 15 days) post-inclusion
  Percentage of patients with at least one adverse event (graded 3 or 4 according to NCI-CTCAE V5.0) at evaluation visit at 3 months.
Frequency of grade 3 - 4 adverse events present at 6 months post-inclusion | At 6 months (± 15 days) post-inclusion
  Percentage of patients with at least one adverse event (graded 3 or 4 according to NCI-CTCAE V5.0) at Follow-up (FU) visit at 6 months.
Percentage of patients with unscheduled hospitalization due to their cancer occurring during the 3 months following inclusion | At 3 months (± 15 days) post-inclusion
  Percentage of patients that required at least one unscheduled hospitalization due to their cancer and/or treatment during the 3 months following their enrollment in the trial based on patient's medical record
Percentage of patients with unscheduled hospitalization due to their cancer occurring during the 6 months following inclusion | At 6 months (± 15 days) post-inclusion
  Percentage of patients that required at least one unscheduled hospitalization due to their cancer during the 6 months following their enrollment in the trial based on patient's medical record
Satisfaction of professionals regarding CONTINUUM+ CONNECT solution and its functioning | Through out the study, up to 10 months. At least once per professional
  Dedicated questionnaire available in French from CONTINUUM+ CONNECT solution
Satisfaction of patients regarding CONTINUUM+ CONNECT solution and its functioning | At 3 months (± 15 days) post-inclusion
  Dedicated questionnaire available in French from CONTINUUM+ CONNECT solution

CONTACTS AND LOCATIONS:
Overall Officials: Philippe BARTHELEMY, MD, Study Chair — Hôpitaux Universitaires de Strasbourg
Locations (13):
- France (13):
  - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy, De
  - Sainte-Catherine, Institut du Cancer Avignon-Provence, Avignon
  - Polyclinique de Blois, Blois
  - Pôle Santé République, Clermont-Ferrand
  - centre Georges François Leclerc, Dijon
  - Chu Dupuytren, Limoges
  - Centre Hospitalier de Morlaix, Morlaix
  - Centre d'oncologie de Gentilly, Nancy
  - Hôpitla privé des Côtes d'Armor - Centre CARIO-HPCA, Plérin
  - Institut Jean Godinot, Reims
  - CHU de Saint-Etienne, Saint-Priest-en-Jarez
  - Centre Paul Strauss, Strasbourg
  - Hôpitaux Universitaires de Strasbourg, Strasbourg